CLINICAL TRIAL: NCT01855178
Title: Pediatric Seizure Alarm: A Pilot Study to Establish Efficacy Parameters
Brief Title: Pediatric Seizure Movement Bed Alarm
Acronym: PedsBedAlarm
Status: Completed | Type: Observational
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, James W. Wheless, Principal Investigator, Le Bonheur Children's Hospital
Other Study IDs: 10-00895-XP
Record Dates: First submitted 2012-02-23; First posted 2013-05-16 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Seizures; Sleep; Epilepsy
Keywords: nocturnal; epilepsy
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Emfit Movement Monitor — Factory settings
  Other Names: control unit D2090; under mattress sensor L-4060SL; Seat sensor L3030SL

SUMMARY:
Nocturnal seizure and Sudden unexplained death in epilepsy patients (SUDEP) are major concerns for parents and creates anxiety and poor sleep conditions for many families dealing with epilepsy. An accurate and reliable system for alerting parents to ongoing seizure activity could make a substantial impact in quality of life and possibly reduce the mortality of epilepsy. No previous studies in the pediatric population have been performed to evaluate this type of monitoring for seizure activity. This is one of the most common questions parents ask in clinic, "Are there any alarms that can tell me when my child is having a seizure at night?" Currently the answer is no. This study has the capability to give us data that may change this answer to yes.

DETAILED DESCRIPTION:
For parents of children with epilepsy, seizures occurring in sleep are a major concern. This frequently leads to many nights of lost sleep for parents and also to unfavorable sleeping arrangements, especially for older children and adolescents. Sudden unexplained death in epilepsy patients (SUDEP) is also a major concern for both parents and neurology practitioners. Patients with epilepsy have increased risk of sudden unexplained death compared to the rest of the population. The risk of sudden death in epilepsy is estimated at 24 times the risk of the general population. Specific risk factors for sudden death have been evaluated and the most frequently reported risk factors include: nocturnal seizures, being in bed, and history of generalized tonic -clonic seizures. Interestingly, one case-control study observed a decreased risk of SUDEP with nighttime monitoring or supervision which raises the possibility that some cases of SUDEP may be preventable if another person is able to give assistance. This finding may indicate that some of these deaths may be preventable if a caregiver could be alerted to seizure activity. Use of "baby monitors", apnea monitors and pulse oximeters to monitor their children at night has been attempted by families; however, these devices are not specific to seizure activity and in the case of apnea monitors and pulse oximeters have frequent false alarms leading to further anxiety and sleep disturbance for families. Therefore, there is a need for a product that can reliably detect seizure activity without such frequent false positives as to interfere with sleep and functional life.

ELIGIBILITY:
Inclusion Criteria:

* epilepsy

Exclusion Criteria:

* non-epileptic

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 200 children and young adults will be enrolled in the study. Patients will be recruited from the population of children and young adults being admitted to the Epilepsy Monitoring Unit at LeBonheur Children's Hospital for evaluation of ongoing seizure disorders.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of nocturnal seizure bed alarm | 5 years
  Measure the occurrence rate of false alarms. Determine if setting parameters for detection can be established according to age and body weight of child/adult.

SECONDARY OUTCOMES:
Measure seizure types best detected using seizure bed alarm system | 5 years
  Determine which seizure types are best detected using the bed alarm system i.e. generalized tonic-clonic, tonic, focal clonic, complex-partial, seizure events.

CONTACTS AND LOCATIONS:
Overall Officials: James W Wheless, MD, Principal Investigator — LeBonheur Children's Hospital
Locations (1):
- LeBonheur Children's Medical Center, Memphis, Tennessee, United States

REFERENCES:
- [Background] Rauhala E, Virkkala J, Himanen SL. Periodic limb movement screening as an additional feature of Emfit sensor in sleep-disordered breathing studies. J Neurosci Methods. 2009 Mar 30;178(1):157-61. doi: 10.1016/j.jneumeth.2008.11.019. Epub 2008 Dec 3. PMID 19100767